CLINICAL TRIAL: NCT04153513
Title: Comparison of the Effect of Lanolin and Breastmilk in the Treatment of Sore and Damaged Nipples in Breastfeeding Women- a Randomized Controlled Trial
Brief Title: Effect of Lanolin and Breastmilk in the Treatment of Sore and Damaged Nipples in Breastfeeding Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Mostar (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Olivera Perić, Olivera Perić MSc, Head nurse Department of Gynecology and Obstetrics, University of Mostar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Study 2
Record Dates: First submitted 2019-09-26; First posted 2019-11-06 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Lanolin; Milk

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will be randomly assigned to two study groups. An envelope containing a note, "mother's milk group" or "lanolin group" will be randomly distributed among women by a midwife who is not a part of the study. The participants will know which group they belong to. A single blind masking will be used during telephone data collection on day three and seven of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lanolin (Experimental)
  Interventions: Drug: Lanolin
- Mother's milk (Active Comparator)
  Interventions: Other: Mother's milk

INTERVENTIONS:
Drug: Lanolin — Lanolin will be applied by hand in a thin layer to the nipple and areola after every breast feed (approximately every 2 to 3 hours) for a maximum of 7 days or until the symptoms of pain and signs of nipple damage have ceased (if noted before 7 days).
  Arms: Lanolin
Other: Mother's milk — After each breast feed (approximately every 2 to 3 hours), a few drops of breast milk will be applyed to the nipple and areola by hand and allow them to air dry. The treatment will last for up to 7 days or until the symptoms of pain and signs of nipple damage have ceased (if noted before 7 days).
  Arms: Mother's milk

SUMMARY:
A randomized controlled study will be conducted at the accredited Baby Friendly Hospital in Mostar, Bosnia and Herzegovina. The study will include primiparas who have established breast feeding at the maternity ward and developed symptoms of painful and sore nipples within 72 hours from childbirth. Participants will be allocated in two groups and will receive education prior to the study.

DETAILED DESCRIPTION:
Recent studies show that early termination of breastfeeding is often associated with painful and sore nipples. Although health professionals recommend various treatments for painful and sore nipples, including alternative treatments, there is currently not enough evidence to recommend specific treatment of painful and sore nipples in lactating women. The primary objective of this study is to compare the effect of lanolin administration and the application of breast milk on the intensity of pain and healing of damaged nipples during breastfeeding. Subjects in the lanolin group will apply lanolin on each nipple and areola after each feeding while subjects in the breast milk group will apply several drops of milk on the nipple after each feed and allow them to air dry. In both groups, the treatment will last for 7 days or until the symptoms of pain and nipple damage have ceased. The main outcome measure is pain, which will be assessed through three time points and will be measured using an abridged version of the McGill Pain Questionnaire. Nipple damage will be assessed by means of a validated assessment tool, the Nipple trauma score. Secondary outcome measures will include breastfeeding efficacy, duration of any/exclusive breastfeeding, reasons for stopping breastfeeding and satisfaction with proposed treatment.The contribution of this study will be reflected in efficient treatment, better care of health professional in the prevention and treatment of damaged and sore nipples, and the study will also contribute in defining the guidelines for the development of procedure in midwifery practice for the treatment of painful and damaged nipples.

ELIGIBILITY:
Inclusion Criteria:

* Primiparas who have given birth to infants born at full term at between 37-41 weeks gestation
* Mothers complaint of nipple pain with any sign of nipple trauma to one or both nipples,
* Access to telephone
* Signed Informed consent

Exclusion Criteria:

* Primiparas with mental disorders
* Mothers allergy to lanolin
* Mothers with abnormal nipples
* Breast hypoplasia
* Infant with cleft palate
* Ankyloglossia
* Unsigned Informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in nipple pain severity | baseline, 3 and 7 days post randomization
  An abbreviated version of the McGill Questionnaire (SF-MPQ) will be used to assess the intensity of nipple pain. For the assessment of the current intensity of pain in the nipples will be used subcategories SF-MPQ, the current assessment of pain (PPI). It consists of a verbal scoring scale with values from 0 to 5, 0= No pain, 1= Mild, 2 = Discomforting, 3= Distressing, 4= Horrible, 5= Excruciating
Nipple damage change | baseline, 3 and 7 days post randomization
  The baseline assessment of nipple damage will be performed by a validated Nipple Trauma Score (NST). The assessment is performed on scales from 0 to 5 where 0 = no macroscopically visible changes in the skin, 1 = erythema or edema or a combination of both, 2 = superficial damage or no scab on <25% of the nipple surface, 3 = superficial damage with or without scab on> 25% of nipple surface, 4 = partial thickness wound with or without scab on <25% of nipple surface, 5 = partial thickness with or without scab on> 25% of nipple surface.
  Three and 7 days after applying the treatment, the condition of the nipple will be evaluated with a Questionnaire on Pain and Damage to the Nipple, where a telephone survey will be performed by the Principal Investigator in order to describe and compare the condition of the nipples.

SECONDARY OUTCOMES:
Assessment of breastfeeding self-efficacy | baseline, 3 and 7 days post randomization
  Breastfeeding self-efficacy will be evaluated by a validated version of the Self-Efficacy Scale-Short Form (BSES-SF). The scale consists of 14 items, with the offered five statements on the Likert scale, from strongly disagree to strongly agree. The sum of grades ranges from 14 to 70, the higher the sum the greater the efficiency of breastfeeding.
Breastfeeding duration and exclusivity. | 3 and 7 days post randomization, 3 and 6 months postpartum
  The way of feeding of the baby in the last 24 hours will be evaluated by the World Health Organization (WHO) breastfeeding categories. The assessment will be conducted through a telephone interview with her mother.
Satisfaction with proposed treatment | 3 and 6 months postpartum
  The evaluation will be conducted by telephone interview with the Maternal Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Olivera Perić, VII, Principal Investigator — Department of Gynecology and Obstetrics, University Clinical Hospital Mostar; Anita Pavičić Bošnjak, VII, Study Chair — Clinical Hospital Centre Zagreb; Vajdana Tomić, VII, Study Chair — Department of Gynecology and Obstetrics, University Clinical Hospital Mostar
Locations (1):
- Department of Gynecology and Obstetrics, University Clinical Hospital Mostar, Mostar, HNŽ, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Result] Pavicic Bosnjak A, Rumboldt M, Stanojevic M, Dennis CL. Psychometric assessment of the croatian version of the breastfeeding self-efficacy scale-short form. J Hum Lact. 2012 Nov;28(4):565-9. doi: 10.1177/0890334412456240. Epub 2012 Sep 6. PMID 22956741
- [Result] Abou-Dakn M, Fluhr JW, Gensch M, Wockel A. Positive effect of HPA lanolin versus expressed breastmilk on painful and damaged nipples during lactation. Skin Pharmacol Physiol. 2011;24(1):27-35. doi: 10.1159/000318228. Epub 2010 Aug 18. PMID 20720454
- [Derived] Peric O, Pavicic Bosnjak A, Mabic M, Tomic V. Comparison of Lanolin and Human Milk Treatment of Painful and Damaged Nipples: A Randomized Control Trial. J Hum Lact. 2023 May;39(2):236-244. doi: 10.1177/08903344221135793. Epub 2022 Nov 18. PMID 36401521
- See also: A Randomized Controlled Trial Evaluating Lanolin for the Treatment of Nipple Pain Among Breastfeeding Women — http://tspace.library.utoronto.ca/bitstream/1807/65631/3/Allen_Kim_201406_PhD_thesis.pdf